CLINICAL TRIAL: NCT06473285
Title: Effects of Esketamine on Consciousness-related Brain Network Characteristics in Patients With Prolonged Disorders of Consciousness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Head of anesthesiology, Principal Investigator, Clinical Professor, Beijing Tiantan Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: LY20240424
Record Dates: First submitted 2024-05-27; First posted 2024-06-25 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Prolonged Disorders of Consciousness
Keywords: Esketamine; Multichannel electroencephalogram; Event-related potential; Brain network characteristics
MeSH Terms: interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy brain volunteers (Active Comparator)
  Interventions: Drug: Drug: Esketamine (Continuous infusion)
- Patients with prolonged disorders of consciousness (Experimental)
  Interventions: Drug: Drug: Esketamine (Continuous infusion)

INTERVENTIONS:
Drug: Drug: Esketamine (Continuous infusion) — Continuous intravenous infusion of ketamine at a dose of 0.3mg/(kg · h). Collect resting state EEG and auditory event-related potential (ERP) before administration (baseline), 60 minutes after administration, 30 and 60 minutes after discontinuation.

SUMMARY:
Prolonged disorders of consciousness (pDoC) are pathologies in which there is a loss of consciousness for more than 28 days. The number of patients with pDoC is increasing as the level of critical care treatment and monitoring improves. However, clinical trials for patients with pDoC are limited by small sample sizes, lack of placebo groups, and use of heterogeneous outcome measures. As a result, few therapies have strong evidence to support their use. In recent years, ketamine has been used with remarkable success in the treatment of neuropsychiatric disorders by inducing neuroplasticity, increasing neurophysiologic complexity, and expanding functional brain connectivity states. Considering increased brain plasticity as well as brain complexity, it may be beneficial for consciousness recovery. In this study, the investigators aimed to explore the effects of esketamine on brain networks and level of consciousness in patients with pDoC, and to discuss its possible use as a wakefulness-promoting treatment for patients with pDoC.

ELIGIBILITY:
Patients with prolonged disorders of consciousness:

Inclusion Criteria:

* Age 18 - 65 years old, native Chinese speaker, dextromanual;
* Chronic disorder of consciousness;
* Spinal cord electrical stimulator implantation under general anesthesia;
* Signed informed consent.

Exclusion Criteria:

* Continuous sedation was administered within 72 hours prior to the study;
* Open head injury, parenchymal resection and other damage of brain structural integrity;
* The intracranial compliance decreased due to hydrocephalus and swelling;
* Known hearing impairment;
* Airway stenosis and various causes of severe ventilation or ventilation dysfunction;
* Known or suspected severe cardiac, pulmonary, hepatic, and renal dysfunction;
* History of drug allergy to esketamine;
* Associated with other mental or neurological diseases;
* Other reasons are not suitable to participate in this study.

Healthy brain volunteers:

Inclusion Criteria:

* Age 18 - 65 years old;
* Patients undergoing surgical treatment under elective general anaesthesia;
* American Society of Anesthesiologists (ASA) I-II;
* Native Chinese speaker;
* Dextromanual;
* Signed informed consent.

Exclusion Criteria:

* Previous history of craniocerebral disease, imaging suggests organic brain lesions;
* People with uncontrolled hypertension, hyperthyroidism, elevated intracranial pressure, epileptic seizures;
* History of drug allergy to esketamine;
* Hearing abnormality;
* History of drug and alcohol abuse;
* People with mental and behavioral disorders.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Entropy index. | During the trial(up to 3 hours for each subject).
  A higher entropy index indicates a higher brain complexity.
Lempel Ziv complexity. | During the trial(up to 3 hours for each subject).
  Higher Lempel Ziv complexity indicates higher brain complexity.

SECONDARY OUTCOMES:
EEG Spectral Characteristics | During the trial(up to 3 hours for each subject).
  EEG power spectrum characteristics of pDoC patients under esketamine. administration, including the δ, θ, α, β, and γ frequency bands.
Cortical Connectivity | During the trial(up to 3 hours for each subject.
  Characteristics of the weighted phase lag index(WPLI) in patients with pDoC. 0 ≤ WPLI ≤ 1, where 0 represents asynchronous and 1 represents synchronous.
Rate of patients recovered consciousness after surgery | During the trial(through study completion, 180 days).
  Rate of patients recovered consciousness 30 days, 90 days, 180 days after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China